CLINICAL TRIAL: NCT01093690
Title: Randomized, Placebo-controlled Trial of Ondansetron Plus Dexamethasone With or Without Metoclopramide as Antiemetic Prophylaxis in Patients Receiving High Dose Cisplatin in Routine Medical Practice
Brief Title: Ondansetron Plus Dexamethasone With or Without Metoclopramide as Antiemetic Prophylaxis After Receiving Cisplatin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Suthinee Ithimakin, Division of medical oncology, department of medicine, Faculty of Medicine Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Si094/2009
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Cancer
Keywords: chemotherapy induced nausea and vomiting, metoclopramide
MeSH Terms: conditions — Neoplasms; Vomiting | interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- metoclopramide (Experimental): ondansetron 8 mg orally twice a day on days 2-5 and dexamethasone 8 mg orally twice a day on days 2-4 plus metoclopramide 20 mg orally four times a day on day 2-5
  Interventions: Drug: metoclopramide
- placebo (Placebo Comparator): ondansetron 8 mg orally twice a day on days 2-5 and dexamethasone 8 mg orally twice a day on days 2-4 plus placebo 20 mg oral four times a day on day 2-5
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: metoclopramide — ondansetron 8 mg orally twice a day on days 2-5 and dexamethasone 8 mg orally twice a day on days 2-4 plus metoclopramide 20 mg oral four times a day on day 2-5
  Other Names: plasil
  Arms: metoclopramide
Drug: placebo — ondansetron 8 mg orally twice a day on days 2-5 and dexamethasone 8 mg orally twice a day on days 2-4 plus placebo 20 mg oral four times a day on day 2-5
  Arms: placebo

SUMMARY:
The objective of this study is to assess the efficacy and tolerability of metoclopramide added to standard antiemetic regimen for prophylaxis of cisplatin-induced emesis.

DETAILED DESCRIPTION:
Ondansetron plus dexamethasone are standard emetic prophylactic agents for highly emetogenic chemotherapy. Metoclopramide is a dopamine antagonist, which may enhance efficacy of ondansetron and dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* schedule to receive first cycle of cisplatin > 50 mg/m^2
* pathologically or histologically confirmed solid cancer
* more than 18 years old
* creatinine clearance more than 50 ml/min
* aminotransferase less than 2 times of upper normal limit

Exclusion Criteria:

* pregnant woman
* patients with episode of vomiting within 24 hours prior to chemotherapy session
* gut obstruction
* brain metastasis
* abdominal or pelvic irradiation
* no history of allergy to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suthinee Ithimakin, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Division of medical oncology, department of medicine Siriraj Hospital, Bangkok, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from April 2009-June 2010.
Pre-assignment Details: All recruited patients were participate enrollment.
Groups:
- Placebo: ondansetron 8 mg twice a day on days 2-5, dexamethasone 8 mg twice a day on days 2-4 plus placebo 20 mg four times a day on day 2-5
Period: Overall Study
Arm/Group | Metoclopramide | Placebo
Started | 83 | 79
Completed | 83 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoclopramide | Placebo | Total
Number analyzed (Participants) | 83 | 79 | 162
Age, Customized [Number; unit: participants]
  Between 18 and 50 years | 41 | 38 | 79
  >= 50 years | 42 | 41 | 83
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 60 | 58 | 118
Region of Enrollment [Number; unit: participants]
  Thailand | 83 | 79 | 162

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Had Complete Response
Description: number of patients who experience no emesis and need no rescue treatment in 5-day period
Time Frame: 5 days after receiving chemotherapy
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Metoclopramide | Placebo
Number analyzed (Participants) | 83 | 79
participants | 50 | 42
Statistical Analysis 1: Comparison: Metoclopramide vs Placebo; the study had 80 percent power to detect an absolute difference of 20 percent in complete response (70% for metoclopramide group vs 50% for control group); Test type: Superiority or Other; p = 0.41, Chi-squared — No adjustment; 1-sided test

2. Secondary Outcome: Toxicities and Severity of Nausea and Vomiting
Time Frame: 5 days after receiving chemotherapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Metoclopramide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/79
Other Adverse Events (participants affected / at risk) | 67/83 | 62/79
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoclopramide (N=83) | Placebo (N=79)
fatigue (General disorders) | 41 (41) | 43 (43)
anorexia (General disorders) | 39 (39) | 46 (46)
headache (General disorders) | 5 (5) | 10 (10)
constipation (Gastrointestinal disorders) | 38 (38) | 29 (29)
sleepiness (General disorders) | 10 (10) | 7 (7)
hiccup (General disorders) | 7 (7) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes